CLINICAL TRIAL: NCT06661239
Title: Effect of the Benson Relaxation Technique on Clinical Outcomes of Oncology Patients Admitted to Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Damanhour university
Record Dates: First submitted 2024-10-19; First posted 2024-10-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-06

CONDITIONS: Oncology Patients; Relaxation Program
Keywords: benson relaxation; Oncology/ cancer patients; Clinical outcomes

STUDY DESIGN:
Intervention Model Description: The Benson relaxation consisted of the following steps: (1) Sitting or lying down quietly in a comfortable position; (2) Closing eyes; (3) Deeply relaxing all muscles, beginning at the feet and progressing up to the face. Keeping them relaxed; (4) Breathing through the nose. (5) Maintaining a passive attitude and permitting relaxation to occur at its own pace; (6) Continuing for 15 minutes. When finished, sit quietly for several minutes, at first with eyes closed and later with eyes opened. Do not stand up for a few minutes.
  According to the agreement, the patients in both groups were required to perform the Benson relaxation technique regularly twice daily (morning and evening) for seven days in a row. Each session lasted 15 minutes.
Who Masked: Participant
Masking Description: The studied patients will be masked for the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The benson group (Experimental): Patients who received the intervention
  Interventions: Behavioral: benson relaxation
- Control group (Placebo Comparator): Patients who receive routine care in units
  Interventions: Behavioral: Routine care in unit

INTERVENTIONS:
Behavioral: benson relaxation — The benson relaxation consisted of the following steps: (1) Sitting or lying down quietly in a comfortable position; (2) Closing eyes; (3) Deeply relaxing all muscles, beginning at the feet and progressing up to the face. Keeping them relaxed; (4) Breathing through the nose. (5) Maintaining a passive attitude and permitting relaxation to occur at its own pace; (6) Continuing for 15 minutes. When finished, sit quietly for several minutes, at first with eyes closed and later with eyes opened. Do not stand up for a few minutes.
  According to the agreement, the patients in both groups were required to perform the Benson relaxation technique regularly twice daily (morning and evening) for seven days in a row. Each session lasted 15 minutes
  Arms: The benson group
Behavioral: Routine care in unit — The routine care include in the unit will be delivered to control group
  Arms: Control group

SUMMARY:
The benson Relaxation Technique (BRT), developed by Dr. Herbert Benson, is a method aimed at reducing stress and anxiety through a series of simple steps designed to elicit the "Relaxation Response." This response is a physiological state that counteracts the harmful effects of stress, characterized by decreased heart rate, lower metabolism, and reduced breathing rate

DETAILED DESCRIPTION:
The benson relaxation consisted of the following steps: (1) Sitting or lying down quietly in a comfortable position; (2) Closing eyes; (3) Deeply relaxing all muscles, beginning at the feet and progressing up to the face. Keeping them relaxed; (4) Breathing through the nose. Becoming aware of breathing. Focus on a word, phrase, a short prayer, or only breathing. (6) Continuing for 15 minutes. When finished, sit quietly for several minutes, at first with eyes closed and later with eyes opened. Do not stand up for a few minutes.

According to the agreement, the patients in both groups were required to perform the Benson relaxation technique regularly twice daily (morning and evening) for three days in a row. Each session lasted 15 minutes

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years
* diagnosed with cancer
* alert and able to communicate.

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients with cognitive impairment
* Patient who unable to communicate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | daily for three days
  measure heart rate per min
Blood pressure | daily for three days
  measure blood pressure in mmHg
Respiratory rate | daily for three days
  measure respiratory rate per min
The Rhodes Index of Nausea, Vomiting, and Retching | daily for three days
  It is a self-report tool designed to assess the severity and impact of nausea, vomiting, and retching on patients' 5-point categorical scales, the interval of each category was (maximum possible score/4-1 ) with the score being zero in the "none" category. For example, if the maximum possible score was 32, then, none: 0, mild: 1-8, moderate: 9-16, severe: 17-24, great: 24-32.
The Numeric Pain Rating Scale | daily for three days
  The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours. scale is the most widely used single-dimension assessment scale.The total score is divided into 4 main categories: zero, which indicates no pain; 1-3 grades, which indicates mild pain; 4-6 grades, which indicate moderate pain; and 7-10 grades, which indicate severe pain
Insomnia Severity Index Scale | daily for three days
  The Insomnia Severity Index (ISI) is a widely used self-report questionnaire designed to assess the severity of insomnia. It consists of seven questions, each rated on a scale that reflects the severity of sleep problems experienced over the last two weeks. The total score is calculated by summing the responses to all seven items, with potential scores ranging from 0 to 28.
  Total Score Calculation 0-7: No clinically significant insomnia 8-14: Subthreshold insomnia 15-21: Clinical insomnia (moderate severity) 22-28: Clinical insomnia (severe)

SECONDARY OUTCOMES:
Icu length | an average three months
  How long patient stay in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Damanhūr, Egypt